CLINICAL TRIAL: NCT04022772
Title: Longitudinal Cohort Study of the Effect of an eHealth Support Program on Patient Reported Outcomes of Women With Breast Cancer
Brief Title: Effect of PACK Health Support Program on Patient Reported Outcomes in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0473; NCI-2019-03897 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0473 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Breast Carcinoma; Breast Ductal Carcinoma In Situ; Invasive Breast Carcinoma; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Practice Guidelines as Topic; Standard of Care; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I (PACK Health program) (Experimental): Patients participate in PACK Health program consisting of weekly contact with an assigned health coach via text message, phone call, and email for 3 months. After 3 months, patients continue to be contacted by the health coach at least once monthly for an additional 3 months.
  Interventions: Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Supportive Care
- GROUP II (standard of care) (Active Comparator): Patients receive standard of care support services over 6 months.
  Interventions: Other: Best Practice; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: GROUP II (standard of care)
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Supportive Care — Participate in PACK Health program
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: GROUP I (PACK Health program)

SUMMARY:
This trial studies the effect of an electronic health (eHealth) support program called PACK Health on patient reported health outcomes in patients with breast cancer. PACK Health monitors breast cancer patients' reported side effects and experience of care when receiving chemotherapy. Participating in the PACK Health coaching program may improve quality of life, decrease hospital admissions and improve overall health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of an eHealth coaching program on the self-reported global health of women with breast cancer, as measured by the National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale version (v.) 1.2.

SECONDARY OBJECTIVES:

I. To evaluate the effect of an eHealth coaching program on the symptom experience of women with breast cancer as measured by the MD Anderson Symptom Inventory-Breast (MDASI-Br).

II. To evaluate the effect of an eHealth coaching program on physical and mental health of women diagnosed with breast cancer as measured by the subscales of the PROMIS Global Health Scale v 1.2.

III. To evaluate the effect of an eHealth coaching program on the symptom experience and global health outcomes of women by:

IIIa. Disease stage. IIIb. Active treatment type (i.e. surgery, radiation, chemotherapy, hormonal therapy, immunotherapy or a combination of these methodologies).

IIIc. Time since diagnosis. IV. To evaluate the effect of an eHealth coaching program on the frequency of emergency room visits and hospital admissions for patients receiving treatment in the ambulatory setting.

V. To evaluate the relationship between financial toxicity, as measured by the Consumer Score for Financial Toxicity (COST), and quality of life, as measured by the Functional Assessment of Quality of Life-Breast (FACT-B).

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients participate in PACK Health program consisting of weekly contact with an assigned health coach via text message, phone call, and email for 3 months. After 3 months, patients continue to be contacted by the health coach at least once monthly for an additional 3 months.

GROUP II: Patients receive standard of care support services over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Able to read, speak and consent in English.
* Individuals with a diagnosis of:

  * First time diagnosis of invasive breast cancer,
  * Ductal carcinoma in situ (DCIS),
  * Recurrent breast cancer off all therapy prior to recurrence
* Currently starting or undergoing active treatment
* Internet access via smart phone, tablet, a computer, or another device with the capacity to receive calls, texts, or e-mails, as well as the electronic study assessments.

Exclusion Criteria:

* Male patients (due to the small number of male breast cancer patients treated annually).
* Individuals for whom there is documentation of inability to provide consent in the medical record.
* Patients who were previously enrolled on protocol 2016-0761.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Patient reported outcomes on global physical and mental health | Up to 6 months
  Measured by the National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale version (v.)1.2. PROMIS v1.2 raw scores will be converted to PROMIS v1.2 t-scores prior to any analyses. Because t scores can only be calculated if a participant answers all 10 items, multiple imputation techniques will be used to estimate the values for missing items. Prior to conducting multiple imputation, the data will first be examined to determine whether missing data are missing completely at random (MCAR), missing at random (MAR) or missing not at random (MNAR). Models will be created separately for physical and mental health. Testing will be 2-sided and conducted with a 0.05 level of statistical significance yielding a family wise Type I error rate of 0.10.

SECONDARY OUTCOMES:
Rate of emergency room visits and hospital admissions | From day 1 to day 180
  A generalized linear mixed model using a log link function will be used to model the rate of emergency room visits and hospital admissions by intervention and time. The number of emergency room visits and hospital admissions will be recorded for each subject from day 1 through day 180 and summarized to correspond to inventory assessment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Hacker, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org